CLINICAL TRIAL: NCT05674149
Title: Image Data Collection Using a Multi-spectral Camera for Computer Vision Algorithms Research and Development
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lumenis Be Ltd. (Industry)
Collaborators: Emek Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: LUM-ABU-SMRT-22-04
Record Dates: First submitted 2022-11-25; First posted 2023-01-06 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Vascular Lesion; Pigmented Lesions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multi-Spectral Camera (Other): Multi-Spectral Camera will be used in order to capture images of different skin conditions
  Interventions: Device: camera

INTERVENTIONS:
Device: camera — photographs using multi-spectral camera

SUMMARY:
This is an observational, single-center, open-label photography evaluation. Any patient that arrives for consultation or treatment at the clinic, presenting the required lesions detailed in the protocol can be included.

DETAILED DESCRIPTION:
This is an observational, single-center, open-label photography evaluation. Any patient that arrives for consultation or treatment at the clinic, presenting the required lesions detailed in the protocol can be included.

The specified lesions can be located on any area of the face or body. For consenting subjects at least 5 close-up images of at least one lesion and one reference image (e.g., subject's skin without any lesion) will be obtained using the Multi-spectral SMART camera. An additional reference image of the lesion area will be taken with a regular camera. Optional images may be taken using a dermatoscop

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all the following inclusion criteria to be entered into the study:

Any patient, male or female of at least 18 years old, who is willing to sign an informed consent form and present at least one of the following conditions:

1. Photoaging (type I - III per Glogau classification)- mixed conditions
2. Epidermal pigmentation / Lentigines (age spots, sun spots)
3. Facial rosacea (Erythematotelangiectatic rosacea and papulopustular rosacea)
4. Facial telangiectasia
5. Poikiloderma
6. Seborrheic keratosis
7. Melasma (Chloasma)

Exclusion Criteria:

Any of the following will exclude the subject from the study:

The study is intended to gather image data so, any patient can be included in the study, and no exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2023-06-21 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Images collection | through study completion, up to 4 months
  Images of different skin condition will be collected using multispectral camera

SECONDARY OUTCOMES:
Images data collection | through study completion, up to 4 months
  for each collected image using multispectral camera, skin an lesion attributes will be evaluated by the investigator. the following attribute will be collected: skin type, lesion type, lesion intensity

CONTACTS AND LOCATIONS:
Locations (1):
- Ha'Emek Medical Center, Afula, Israel

IPD SHARING:
Plan to Share IPD: No